CLINICAL TRIAL: NCT00164788
Title: A Randomized Comparison of High Dose Oral to Intravenous Esomeprazole in Patients After Endoscopic Control to Their Bleeding Peptic Ulcers: an Intra-gastric pH Study.
Brief Title: A Comparison of Gastric pH Control With High Dose Intravenous or Oral Esomeprazole
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No suitable patients and many patients refused the study
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ne_pH
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Gastrointestinal Hemorrhage
Keywords: 24 hours pH monitoring
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IV Nexium (Active Comparator): Intravenous bolus injection of esomeprazole (Astra Pharmaceutica AG, Dietikon, Switzerland) 80mg followed by continuous intravenous infusion of 8mg per hour for 24 hours
  Interventions: Drug: Intravenous bolus injection of esomeprazole
- Oral Nexium (Active Comparator): Oral esomeprazole (Astra Pharmaceutica AG, Dietikon, Switzerland) 40mg every 12 hours for 24 hours
  Interventions: Drug: Oral esomeprazole

INTERVENTIONS:
Drug: Intravenous bolus injection of esomeprazole — 80mg followed by continuous intravenous infusion of 8mg per hour for 24 hours
  Other Names: IV Nexium
  Arms: IV Nexium
Drug: Oral esomeprazole — 40mg every 12 hours for 24 hours
  Other Names: Oral Nexium
  Arms: Oral Nexium

SUMMARY:
The investigators hypothesize that high dose esomeprazole 80mg given as a bolus, followed by 8mg/h would render gastric pH near neutral and that pH control with esomeprazole given in such a high dose either intravenous or orally is identical.

DETAILED DESCRIPTION:
Bleeding peptic ulcer is a common and life threatening condition. Endoscopic therapy has become the mainstay of controlling bleeding. Recurrent bleeding after endoscopic control occurs in about 20% of patients with a high associated mortality. We previously demonstrated that the adjunct use of high dose proton pump inhibitor reduces risk of recurrent bleeding and thereby improves patients' outcome [Lau JY N Engl J Med 2000]. The newer PPI, esomeprazole, is an S-isomer of omeprazole. Esomeprazole is more effective in gastric acid control as measured by both basal and pentagastrin acid output when compared to omeprazole. Esomeprazole when given orally at a lower dose achieves a similar gastric control than intravenous esomeprazole. The gastric pH with a high dose esomeprazole when given either orally or intravenously has not been measured among Hong Kong Chinese. If a high dose oral esomeprazole achieves a similar pH control near gastric neutrality, the oral regime can be used in place of the intravenous formulation. This represents significant convenience in dosing and cost savings.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted with diagnosis of upper gastrointestinal bleeding aged between 18 and 80
* Endoscopic confirmation of a bleeding duodenal or gastric ulcer to which endoscopic control has been obtained
* Absence of H. pylori infection
* Informed written consent

Exclusion Criteria:

* Known incompatibility to the study drugs;
* Known incompatibility and hypersensitivity to proton pump inhibitor
* H. pylori infection
* Recent H2RA or PPI use (within last 4 weeks)
* Concomitant use of medications that may interfere gastric acid secretion or motility (e.g. anticholinergic, metoclopramide, domperidone)
* Pregnancy or lactation;
* Non-compliance e.g. mental subordination
* Nasopharyngeal or oropharyngeal pathology that would prevent passage of a nasal catheter
* Significant liver disease as PPI is metabolized by the cytochrome P-450 system
* Previous gastric surgery
* Chronic Aspirin user
* Presence of esophageal/ gastric varices
* Moribund patients, terminal malignancy & patients with severe renal disease
* Patient unable to give written consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
The primary measure of this study is the median gastric pH over 24-hour monitoring. | 24 hours

SECONDARY OUTCOMES:
acid suppressing activity, notably the rate of onset of action, between the two treatment regimens: 1. Percentage time of pH<6 2. Time to reach pH 6 3. Median gastric pH in the first 6 and 12 hours | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: James YW Lau, MD, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong (sar), China